CLINICAL TRIAL: NCT02343367
Title: Pediatric Obesity Management Intervention Trial for Hispanic Families
Brief Title: Health4Kids Intervention Trial for Hispanic Families
Acronym: H4K
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); The University of Texas at San Antonio (Other); Bexar County Hospital District DBA University Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC20130465H; R01HD075936 (NIH)
Record Dates: First submitted 2015-01-06; First posted 2015-01-22 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Pediatric Obesity
Keywords: Hispanic; overweight; families; pediatric; primary care
MeSH Terms: conditions — Pediatric Obesity; Overweight | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (Active Comparator): Brief patient-centered behavioral counseling using the Healthy Lifestyle Prescription, health education materials and a community resource guide. Follow-up visits scheduled at 1, 6, and 12 months. Parent receives weekly general health education cell phone text messages for 12 months
  Interventions: Behavioral: behavioral counseling; Other: Education Materials; Behavioral: Text messages
- Pediatric Obesity Management (Experimental): All elements of standard care plus a family-based face to face counseling session with a health educator, telephone counseling, mailed newsletters and regularly scheduled cell phone text messages with tips and motivational messages for healthy eating and PA, as well as information on community events and resources.
  Interventions: Behavioral: behavioral counseling; Other: Education Materials; Behavioral: Face to face counseling session; Behavioral: Text messages; Behavioral: Telephone Counseling; Behavioral: Newsletters

INTERVENTIONS:
Behavioral: behavioral counseling — Pediatrician trained in motivational interviewing techniques provides brief lifestyle behavioral counseling to child and parent using a Healthy Lifestyle Prescription
Other: Education Materials — Health education materials about healthy eating and physical activity and a community resource guide
Behavioral: Face to face counseling session — 30 minute face-to-face family-centered behavioral counseling session delivered by a health educator
  Arms: Pediatric Obesity Management
Behavioral: Text messages — regularly scheduled cell phone text messages for 12 months
  Other Names: SMS
Behavioral: Telephone Counseling — 14 telephone counseling sessions delivered by a health educator using motivational interviewing techniques. Two sessions per month for the first two months followed by one session per month for 10 months
  Arms: Pediatric Obesity Management
Behavioral: Newsletters — 12 monthly newsletters mailed to participant homes
  Arms: Pediatric Obesity Management

SUMMARY:
The H4K Trial is a randomized controlled trial to improve children's body composition by testing a comprehensive, culturally and linguistically relevant, family-oriented intervention for overweight and obese Hispanic children (ages 6-11) in three pediatric clinics in San Antonio, Texas. The H4K trial will test the efficacy of a 6-month pediatric obesity management intervention (physician counseling plus telephone counseling, newsletters and text messages) compared to standard care (physician counseling only) on three outcomes: 1) body composition (i.e., waist circumference, weight and z-BMI); 2) insulin, glucose and cholesterol levels; and 3) behavior change in physical activity (PA), sedentary behavior and consumption of sugary beverages and fruits and vegetables. The investigators will recruit 230 overweight and obese children-and a parent or guardian for each-and randomize them to the H4K intervention (n = 115 child/parent dyads) or standard care (n = 115 child/parent dyads). The investigators hypothesize that intervention children will significantly improve their body composition, increased their PA levels and diet quality (more fruits and vegetables and less sugary beverages), and decrease their sedentary activity, compared to children in standard care. If successful, this study will generate new scientific knowledge about effective Hispanic family-based approaches for obesity prevention with high potential for replication in underserved areas across the nation.

DETAILED DESCRIPTION:
Given the continuing rise of the U.S. Hispanic population, reversing the Hispanic childhood obesity epidemic is critical to the nation's future health. Mexican American children and those from socioeconomically disadvantaged families often are far more overweight and obese than their peers, heightening their risk for obesity-related health complications. Our proposed randomized controlled trial, the Health4Kids (H4K) Trial for Hispanic Families, aims to improve Hispanic children's body composition by testing a comprehensive, culturally and linguistically relevant, family-oriented intervention for overweight and obese (body mass index (BMI) between the 85th and 99.9thth (<99th) percentile for age and gender) Hispanic children ages 6-11 in pediatric clinics in San Antonio, Texas, a largely Hispanic city. Our team, formed during our pilot research funded by the Centers for Medicare and Medicaid Services (1H0CMS030457), unites academic investigators and community partners with experience working together to conduct behavioral and clinical interventions and outreach with Hispanics. The H4K trial will test the efficacy of a 6-month pediatric obesity management intervention (physician counseling plus telephone counseling, newsletters and text messages) compared to standard care (physician counseling only) on three outcomes: 1) body composition (i.e., waist circumference, weight and z-BMI); 2) insulin, glucose and cholesterol levels; and 3) behavior change in physical activity (PA), sedentary behavior and consumption of sugary beverages and fruits and vegetables. We will recruit 230 overweight and obese children-and a parent or guardian for each-and randomize them to the POM intervention (n = 115 child/parent dyads) or standard care (n = 115 child/parent dyads). From a baseline, we will measure the impact of the trial on the primary outcome (body composition) and secondary outcomes (insulin, glucose and cholesterol levels and several specific health behavior changes) at 1 month, 6 and 12 months post-randomization. We also will evaluate the critical role of parenting strategies and changes in the home environment as mediators of intervention effects. We hypothesize that intervention children will significantly improve their body composition, increased their PA levels and diet quality (more fruits and vegetables and less sugary beverages), and decrease their sedentary activity, compared to children in standard care. If successful, this study will generate new scientific knowledge about effective Hispanic family-based approaches for obesity prevention with high potential for replication in underserved areas across the nation.

ELIGIBILITY:
Inclusion Criteria:

* A child is eligible for the POM trial for meeting the following criteria:

  * identified by parent or legal guardian as Hispanic
  * age 6-11
  * overweight or obese (BMI between the 85th and 99.9thth (<99th) percentile for age and gender
  * one parent/guardian that the child resides with full-time must agree to participate in intervention and evaluation activities.

Exclusion Criteria:

* A child will be excluded if he/she has:

  * a mental, emotional, or physical handicap identified by parents or health care provider that may interfere with study participation
  * a diagnosis of cardiovascular, pulmonary, or digestive disease
  * parent without a cell phone
  * parent unable or not willing to receive text messages
  * child or parent planning to move from the local area within the time span of the study.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 518 (Actual)
Dates: Start 2015-01; Primary Completion 2019-11-19 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in weight (kg) | 6 months
  Weight will be measured using a portable Tanita Body Composition Analyzer SC-331S following standard protocol.
Change from baseline in waist circumference (cm) | 6 months
  Waist circumference (minimum waist girth) will be measured to the nearest 0.1 cm using a Myotape tape measure at the midpoint between the right iliac crests and the lower ribs when the subject is standing erect with feet together
Change from baseline in body mass index (BMI z score) | 6 months
  BMI will be calculated as weight (kg)/height squared (m2). Weight will be measured by bioelectrical impedance analysis (BIA) using the foot-to-foot pressure contact electrode BIA technique using a portable Tanita Body Composition Analyzer SC-331S following standard protocol. Height will be measured to the nearest 0.1 inch using a SECA brand stadiometer.

SECONDARY OUTCOMES:
Change from baseline in fasting insulin (µIu/mL) | 6 months
  Fasting samples of serum will be drawn by a phlebotomist and processed by a commercial laboratory.
Change from baseline in fasting glucose (mg/dL) | 6 months
  Fasting samples of serum will be drawn by a phlebotomist and processed by a commercial laboratory.
Change in cholesterol (lipid panel: fasting total cholesterol, HDL cholesterol, LDL cholesterol and triglycerides) from baseline (mg/dL) | 6 months
  Fasting samples of serum will be drawn by a phlebotomist and processed by a commercial laboratory.
Change from baseline in moderate-to-vigorous physical activity (minutes/week) | 6 months
  Minutes per week of MVPA is assessed using accelerometry.
Change from baseline in consumption of sugar-sweetened beverages (servings/week) | 6 months
  Sugar-sweetened beverage consumption is assessed using the Block Kids Food Screener (Last Week version).
Change from baseline in consumption of fruits and vegetables (servings/day) | 6 months
  Fruit and vegetable consumption is assessed using the Block Kids Food Screener (Last Week version).

CONTACTS AND LOCATIONS:
Overall Officials: Deborah M Parra-Medina, PhD, Principal Investigator — UT Health San Antonio
Locations (1):
- University of Texas Health Science Center San Antonio, San Antonio, Texas, United States